CLINICAL TRIAL: NCT05751785
Title: Investigation of the Effectiveness of Shockwave Therapy, Photobiomodulation, and Physical Therapy in the Management of Non-insertional Achilles Tendinopathy
Brief Title: Shockwave, Photobiomodulation, and Physical Therapy for Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Musculoskeletal Injury Rehabilitation Research for Operational Readiness (U.S. Federal Agency)
Collaborators: Fort Belvoir Community Hospital (U.S. Federal Agency); The Geneva Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Photomedicine Project 10
Record Dates: First submitted 2023-01-27; First posted 2023-03-02 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Achilles Tendinopathy
MeSH Terms: interventions — Physical Therapy Modalities; Extracorporeal Shockwave Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Physical Therapy (PT) Only (Active Comparator): Participants in the PT only arm will follow the PT program outlined above. Twice a week for three weeks, a team member will check-in with the participants to ensure physical therapy exercise adherence, and response to treatment. During the second check-in of the week, the study team member will also ensure the participant is keeping their activity/medication/pain log; the study team member will also deliver the DVPRS with supplemental questions. (See Appendix F for Check-in Data Collection CRF). These check-ins may occur virtually or in person.
  In Part 1, the physical therapy only arm requires 8 visits. The participants will complete 2 check-in visits each week (remote or in person), for three weeks. Follow-up data will be collected at 6 weeks (virtual or in-person) and at 3 months (in-person).
  Interventions: Other: Physical Therapy
- PT + Photobiomodulation Therapy (PBMT) (Active Comparator): The physical therapy + photobiomodulation therapy arm will receive PBMT twice a week, for three weeks, in addition to the PT treatment described above.
  A member of the study team will measure the treatment area according to a standard protocol (Appendix N PBM Dose Calculations), to calculate and determine the treatment time, approximately 5-20 minutes. PBMT will be delivered at 25W.
  Interventions: Other: Physical Therapy; Device: Photobiomodulation Therapy
- PT + Shockwave Therapy (SWT) (Active Comparator): The physical therapy + shockwave therapy arm will receive SWT once a week for three weeks in addition to the PT treatment described above. Twice a week, for three weeks, a team member will check-in with the participants to ensure physical therapy exercise adherence, and response to treatment. During the second check-in of the week, the study team member will also ensure the participant is keeping their activity/medication/pain log; the study team member will also deliver the DVPRS with supplemental questions. (See Appendix F for Check- in Data Collection CRF). The first check-in of the week will occur in-person after the SWT, if, however, this is not feasible, it may be conducted virtually; the second check-in of the week may occur virtually or in-person.
  In total, participants will receive one SWT treatment each week (in person) and complete two check-ins each week (remote or in person), for three weeks. The SWT will take approximately 5-20 minutes.
  Interventions: Other: Physical Therapy; Device: Shockwave Therapy
- PT + SWT and PBMT (Active Comparator): The PT + SWT + PBMT arm will receive both SWT and PBMT treatments in addition to PT treatment described above. Participants will receive PBMT twice a week and SWT once a week, for three weeks. The SWT visit may be combined with a PBMT visit in the same week. Up to two times each week after a treatment visit (for three weeks), a team member will check-in with the participants to ensure physical therapy exercise adherence, and response to treatment. During the second check-in of the week, the team member will also ensure the participant is keeping their activity/medication/pain log; the team member will also deliver the DVPRS with supplemental questions. When/if needed, these check-ins may occur virtually. (See Appendix F for check-in data collection CRF).
  In Part 1, the PT+ SWT + PBMT treatment arm requires 8 visits: 3 for PBMT alone with check- ins (in person), 3 for PBMT & SWT with check-ins (in person), 6-week follow-up (virtual or in-person), and 3-month follow-up (in person).
  Interventions: Other: Physical Therapy; Device: Shockwave Therapy; Device: Photobiomodulation Therapy

INTERVENTIONS:
Other: Physical Therapy — All participants may complete a PT program as standard of care (SOC) treatment addressing individual strength, mobility, and flexibility deficits in both proximal (e.g. spine and hip girdle) along with distal (thigh, leg, and foot/ankle) muscle groups. The provider may also use other modalities to address distal issues. To standardize the loading program, all participants will be given an at-home exercise program designed by Dr. Karin Sibernagel for progressive Achilles tendon loading. The participants will also follow the University of Delaware Return to Sport protocol for return to running. This will be completed alongside the standard of care PT participants will be receiving.
  Other Names: SOC PT
Device: Shockwave Therapy — A medical provider will conduct SWT on study participants using the OrthoPlus Ultra 100. This Extracorporeal Pressure Activation Treatment device will be used at a radial shockwave of 3000 counts treatment settings of 15 Hz minimum 2 bars with a focus applicator head at mid-portion of Achilles using clinical focusing technique, and 3000 counts at 15 Hz minimum 2.5 bars using broad oscillator to myotendinous region and over symptomatic areas of gastrocnemius and soleus, treatment will be applied distally to proximally to facilitate lymphatic return adjusting treatment air pressure and amount of force applied by applicator head by patient comfort. The maximum setting for each treatment applicator will be 4 bars of air pressure, and the first 500 counts using each applicator will be applied at 1.5 bars to help desensitize the tissue prior to increasing energy settings. The settings used for each participant will be recorded and followed in a similar approach to treatment.
  Other Names: SWT
  Arms: PT + SWT and PBMT; PT + Shockwave Therapy (SWT)
Device: Photobiomodulation Therapy — PBMT is delivered with the LightForce® XPi 25W device through the Smart Hand Piece technology. The therapy is transmitted with a rolling glass massage ball at 10 Joules/cm^2 that is applied in a serpentine manner over the site of injury.
  Other Names: PBMT
  Arms: PT + Photobiomodulation Therapy (PBMT); PT + SWT and PBMT

SUMMARY:
The goal of this clinical trial is to learn more about and compare the effectiveness of standard of care (SOC) physical therapy (PT), PT with photobiomodulation therapy (PBMT; low-level laser therapy), PT with shockwave therapy (SWT; high-energy acoustic wave therapy), and PT with PBMT and SWT, to improve function, decrease pain, and resolve symptoms in individuals with non-insertional Achilles tendinopathy. The main question it aims to answer is:

• What is the most effective treatment method for non-insertional Achilles tendinopathy?

Participants will

Researchers will compare PT, PT + SWT, PT + SWT and PBMT to assess the most effective treatment for Achilles tendinopathy.

DETAILED DESCRIPTION:
Non-insertional Achilles Tendinopathy (AT) is a common overuse injury in adults who are both athletes and nonactive. Tendinopathy occurs when there is either a failed healing response or the failure of normal turnover or remodeling response, and results in pain and limited movement. In the military, lower-extremity injuries due to overuse, (e.g., AT) are the most common category of injuries. The most common treatment of choice for AT is exercise loading programs, however eccentric strengthening (ECC) may only improve symptoms in approximately 60% of patients. Laser-induced photobiomodulation (PBM) has been shown to increase cell proliferation and metabolism, which may aid in the repair and remodeling process. Studies have found that PBM was effective in the treatment of AT. Extracorporeal shockwave therapy (ESWT) is a process in which energy is delivered to the muscles or tendons for pain relief. Current literature supports the use of ESWT as an effective treatment for AT in combination with ECC. Overall, studies indicate that ESWT and photobiomodulation therapy (PBMT) will be effective in treating tendon injuries such as AT, however, these treatment methods have not been evaluated in comparison or combination with each other. The sub-section of AT amongst Active-Duty personnel has very limited research and given the high prevalence, should be addressed. Therefore, our study will compare three different treatment arms utilizing traditional physical therapy (PT), PT plus ESWT, PT plus PBMT, and PT plus ESWT and PBMT. Both self-reported questionnaires and measured outcomes will be used to assess the most effective treatment for AT.

ELIGIBILITY:
Inclusion Criteria:

* DEERS Eligible
* Between the ages of 18-64
* Currently Active Duty in any of the US Armed Forces
* Clinical diagnosis of mid-portion Achilles tendinopathy (including both unilateral and bilateral) by a healthcare provider based on accepted diagnostic criteria.
* Able to read and understand English language for consent purposes
* Able to commit to 3-weeks of intervention and 6-months of follow-up

Exclusion Criteria:

* Primary insertional Achilles tendinopathy
* Platelet Rich Plasma (PRP), corticosteroid injection, or prolotherapy within 3 months
* Received dry needling within the past 4 weeks
* Previously completed the Silbernagel protocol for Achilles tendinopathy within the past 3 months
* Received SWT within the past 3 months to their Achilles
* Tattoo in the area of treatment (due to sensitivity to PBMT)
* Current use of pacemaker
* Patients with a known underlying cardiac disease that could be affected by SWT
* Patients with neuropathy affecting sensation to pain
* Current use of medications associated with sensitivity to heat or light (e.g. amiodarone, chlorpromazine, doxycycline, hydrochlorothiazide, nalidixic acid, naproxen, piroxicam, tetracycline, thioridazine, voriconazole)
* Current or chronic sciatica (lumbosacral radiculopathy) resulting in chronic or intermittent lower extremity pain, numbness, or tingling.
* Achilles tendon tear or prior Achilles tendon surgery
* Recent lower extremity injury within the last 3 months that required professional medical attention (e.g., ankle sprain, meniscus)
* Concurrent participation in another research study addressing pain issue
* Previously enrolled in the study for contralateral (opposite) leg
* Currently pregnant or plan to become pregnant during intervention period (safety of PBM not established in pregnancy) as determined by hCG urine test
* Diagnosis of rheumatological disease/connective tissue condition, symptomatic arthritis of foot and ankle, a primary running related injury outside of Achilles tendinopathy, or other contraindications to PBMT or SWT

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy D Schroeder, Principal Investigator — Madigan Army Medical Center
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 48 participants consented to be in the study. However, 2 participants were withdrawn prior to randomization due to failing formal screening criteria. This left 46 participants to be randomized into a study arm assignment.
Pre-assignment Details: Formal Screening (prior to study arm randomization):
  Post-consent, secondary exclusion of pregnancy will be determined by an hCG urine pregnancy test for females of child-bearing age and capacity.
  Additionally, all participants will be screened for insertional AT as the primary clinical diagnosis with a 3 part test. If the insertional AT component is identified as the primary source of Achilles pain, we formally withdrew the participants from the study prior to randomization.
Groups:
- Physical Therapy (PT) Only: In Part 1, the physical therapy only arm requires 8 visits. The participants will complete 2 check-in visits each week (remote or in person), for three weeks. Follow-up data will be collected at 6 weeks (virtual or in-person) and at 3 months (in-person). All participants may complete a PT program as standard of care (SOC) treatment addressing individual strength, mobility, and flexibility deficits in both proximal (e.g. spine and hip girdle) along with distal (thigh, leg, and foot/ankle) muscle groups. The provider may also use other modalities to address distal issues. To standardize the loading program, all participants will be given an at-home exercise program designed by Dr. Karin Sibernagel for progressive Achilles tendon loading. The participants will also follow the University of Delaware Return to Sport protocol for return to running. This will be completed alongside the standard of care PT participants will be receiving.
- PT + Photobiomodulation Therapy (PBMT): The physical therapy + photobiomodulation therapy arm will receive PBMT twice a week, for three weeks, in addition to the PT treatment described above.
  A member of the study team will measure the treatment area according to a standard protocol (Appendix N PBM Dose Calculations), to calculate and determine the treatment time, approximately 5-20 minutes. PBMT will be delivered at 25W.
  Physical Therapy: All participants may complete a PT program as standard of care (SOC) treatment addressing individual strength, mobility, and flexibility deficits in both proximal (e.g. spine and hip girdle) along with distal (thigh, leg, and foot/ankle) muscle groups. The provider may also use other modalities to address distal issues. To standardize the loading program, all participants will be given an at-home exercise program designed by Dr. Karin Sibernagel for progressive Achilles tendon loading. The participants will also follow the University of Delaware Return to Sport protocol for return to running. This will be completed alongside the standard of care PT participants will be receiving.
  Photobiomodulation Therapy: PBMT is delivered with the LightForce® XPi 25W device through the Smart Hand Piece technology. The therapy is transmitted with a rolling glass massage ball at 10 Joules/cm^2 that is applied in a serpentine manner over the site of injury.
- PT + Shockwave Therapy (SWT): The physical therapy + shockwave therapy arm will receive SWT once a week for three weeks in addition to the PT treatment.
  In total, participants will receive one SWT treatment each week (in person) and complete two check-ins each week (remote or in person), for three weeks. The SWT will take approximately 5-20 minutes.
  Shockwave Therapy: A medical provider will conduct SWT on study participants using the OrthoPlus Ultra 100. This Extracorporeal Pressure Activation Treatment device will be used at a radial shockwave of 3000 counts treatment settings of 15 Hz minimum 2 bars with a focus applicator head at mid-portion of Achilles using clinical focusing technique, and 3000 counts at 15 Hz minimum 2.5 bars using broad oscillator to myotendinous region and over symptomatic areas of gastrocnemius and soleus, treatment will be applied distally to proximally to facilitate lymphatic return adjusting treatment air pressure and amount of force applied by applicator head by patient comfort. The maximum setting for each treatment applicator will be 4 bars of air pressure, and the first 500 counts using each applicator will be applied at 1.5 bars to help desensitize the tissue prior to increasing energy settings. The settings used for each participant will be recorded and followed in a similar approach to treatment.
- PT + SWT and PBMT: The PT + SWT + PBMT arm will receive both SWT and PBMT treatments in addition to PT treatment described. Participants will receive PBMT twice a week and SWT once a week, for three weeks. The SWT visit may be combined with a PBMT visit in the same week. Up to two times each week after a treatment visit (for three weeks), a team member will check-in with the participants to ensure physical therapy exercise adherence, and response to treatment. During the second check-in of the week, the team member will also ensure the participant is keeping their activity/medication/pain log; the team member will also deliver the DVPRS with supplemental questions. When/if needed, these check-ins may occur virtually. (See Appendix F for check-in data collection CRF).
  In Part 1, the PT+ SWT + PBMT treatment arm requires 8 visits: 3 for PBMT alone with check- ins (in person), 3 for PBMT & SWT with check-ins (in person), 6-week follow-up (virtual or in-person), and 3-month follow-up (in person).
Period: Baseline to 3-Month Follow-Up
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Started | 11 | 11 | 12 | 12
Completed | 9 | 10 | 11 | 10
Not Completed | 2 | 1 | 1 | 2
Period: 3-Month Follow-Up to End of Study
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Started | 9 | 10 | 11 | 10
Cross-over Treatment: PT Only | 2 | 0 | 0 | 1
Cross-over Treatment: PT+PBMT | 1 | 0 | 2 | 0
Cross-over Treatment: PT+SWT | 1 | 3 | 1 | 1
Cross-over Treatment: PT+SWT+PBMT | 5 | 6 | 6 | 7
Cross-over Treatment: Declined Additional Treatment | 0 | 1 | 1 | 1
Completed | 8 | 9 | 9 (1 participant was lost to follow up prior to them electing a crossover treatment and 1 participant was lost to follow up after electing crossover treatment.) | 10
Not Completed | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT | Total
Number analyzed (Participants) | 11 | 11 | 12 | 12 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 12 | 12 | 46
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 3 | 11
  Male | 9 | 9 | 8 | 9 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White (not Hispanic | 6 | 7 | 5 | 5 | 23
  Race/Ethnicity: Asian or Pacific Islander | 2 | 0 | 0 | 2 | 4
  Race/Ethnicity: Black or African American (not Hispanic) | 3 | 3 | 3 | 2 | 11
  Race/Ethnicity: American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Race/Ethnicity: Hispanic | 0 | 0 | 4 | 3 | 7
  Race/Ethnicity: Other | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 12 | 12 | 46

OUTCOME MEASURES:

1. Primary Outcome: Victorian Institute of Sports Assessment - Achilles (VISA-A)
Description: The VISA-A (Victorian Institute of Sport Assessment - Achilles) is a questionnaire designed to assess the severity of Achilles tendinopathy. It consists of eight questions that evaluate pain, function in daily life, and sports activities. The minimum score is 0 and the maximum score is 100, with lower scores indicating more severe symptoms and limitations
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 11 | 11 | 12 | 12
score on a scale | 37.55 (15.56) | 43.82 (18.88) | 36.08 (20.55) | 46.92 (13.17)

2. Primary Outcome: Victorian Institute of Sports Assessment - Achilles (VISA-A)
Description: as for outcome 1
Time Frame: 3-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 12 | 10
score on a scale | 56.33 (19.86) | 63.90 (12.91) | 50.17 (16.92) | 58.30 (18.25)

3. Primary Outcome: Victorian Institute of Sports Assessment - Achilles (VISA-A)
Description: as for outcome 1
Time Frame: 6-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 9 | 11 | 10
score on a scale | 61.11 (23.80) | 64 (14.75) | 54.09 (17.35) | 63.20 (19.59)

4. Primary Outcome: Victorian Institute of Sports Assessment - Achilles (VISA-A)
Description: as for outcome 1
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 09 | 10 | 11 | 10
score on a scale | 69.33 (17.67) | 61.10 (20.63) | 58.10 (16.21) | 68.40 (15.90)

5. Primary Outcome: Victorian Institute of Sports Assessment - Achilles (VISA-A)
Description: as for outcome 1
Time Frame: 6-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 8 | 9 | 9 | 10
score on a scale | 67.50 (19.51) | 76.11 (20.37) | 61.22 (18.21) | 69 (18.99)

6. Primary Outcome: Lower Extremity Functional Scale (LEFS)
Description: The Lower Extremity Functional Scale (LEFS) is a questionnaire used to assess a person's ability to perform everyday activities involving the lower limbs. It consists of 20 questions, each scored from 0 to 4, with a minimum score of 0 and maximum total score of 80.
  Key Points: Higher scores indicate better lower extremity function. Lower scores suggest greater disability or difficulty in movement.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 11 | 11 | 12 | 12
score on a scale | 47.91 (14.47) | 50.10 (19.64) | 46.75 (16.87) | 59.55 (12.90)

7. Primary Outcome: Lower Extremity Functional Scale (LEFS)
Description: as for outcome 6
Time Frame: 3-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 12 | 10
score on a scale | 51.33 (18.76) | 60.90 (19) | 47.75 (17.58) | 57.70 (17.60)

8. Primary Outcome: Lower Extremity Functional Scale (LEFS)
Description: as for outcome 6
Time Frame: 6-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 9 | 11 | 10
score on a scale | 60.78 (12.60) | 62.11 (15.71) | 55.27 (14.43) | 64.30 (9.68)

9. Primary Outcome: Lower Extremity Functional Scale (LEFS)
Description: as for outcome 6
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 09 | 10 | 11 | 10
score on a scale | 65.11 (14.47) | 65.30 (15.30) | 54.10 (18.18) | 60.40 (18.58)

10. Primary Outcome: Lower Extremity Functional Scale (LEFS)
Description: as for outcome 6
Time Frame: 6-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 8 | 9 | 9 | 10
score on a scale | 62.38 (17.09) | 64.89 (19.14) | 62.33 (15.53) | 67.10 (10.94)

11. Primary Outcome: Defense and Veteran's Pain Rating Scale (DVPRS)
Description: The Defense and Veterans Pain Rating Scale (DVPRS) is a pain assessment tool designed specifically for military personnel and veterans Rating scale from 0-10. Higher scores equal worse outcomes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 11 | 11 | 12 | 12
score on a scale | 4.27 (1.66) | 3.50 (2.87) | 5.58 (2.29) | 3.27 (1.96)

12. Primary Outcome: Defense and Veteran's Pain Rating Scale (DVPRS)
Description: as for outcome 11
Time Frame: 3-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 12 | 10
score on a scale | 2.67 (1.33) | 2.50 (2.50) | 4.17 (2.15) | 2.60 (1.80)

13. Primary Outcome: Defense and Veteran's Pain Rating Scale (DVPRS)
Description: as for outcome 11
Time Frame: 6-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 09 | 09 | 11 | 10
score on a scale | 2.33 (1.83) | 2.22 (1.93) | 3.64 (2.84) | 1.80 (1.72)

14. Primary Outcome: Defense and Veteran's Pain Rating Scale (DVPRS)
Description: as for outcome 11
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 11 | 10
score on a scale | 1.89 (1.91) | 2.30 (2.65) | 2.80 (2.04) | 2.00 (1.84)

15. Primary Outcome: Defense and Veteran's Pain Rating Scale (DVPRS)
Description: as for outcome 11
Time Frame: 6-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 08 | 09 | 09 | 10
score on a scale | 1.88 (1.90) | 1.67 (2.00) | 2.11 (2.47) | 2.60 (2.65)

16. Primary Outcome: University of Wisconsin Running Injury and Recovery Index (UWRI)
Description: The University of Wisconsin Running Injury and Recovery Index (UWRI) is a questionnaire designed to assess a runner's recovery from running-related injuries. Scores range from 0-36, with higher scores equaling better outcomes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 11 | 11 | 12 | 12
score on a scale | 9.91 (6.24) | 12 (5.88) | 12 (7) | 12.18 (7.57)

17. Primary Outcome: University of Wisconsin Running Injury and Recovery Index (UWRI)
Description: as for outcome 16
Time Frame: 3-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 12 | 10
score on a scale | 15.56 (4.69) | 14.90 (7.12) | 13.42 (9.38) | 14.10 (8.17)

18. Primary Outcome: University of Wisconsin Running Injury and Recovery Index (UWRI)
Description: as for outcome 16
Time Frame: 6-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 9 | 11 | 10
score on a scale | 16.11 (6.64) | 16.44 (8) | 13.36 (8.05) | 16.40 (8.09)

19. Primary Outcome: University of Wisconsin Running Injury and Recovery Index (UWRI)
Description: as for outcome 16
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 11 | 10
score on a scale | 17.89 (4.95) | 17.30 (7.40) | 15.50 (6.99) | 20.80 (7.07)

20. Primary Outcome: University of Wisconsin Running Injury and Recovery Index (UWRI)
Description: as for outcome 16
Time Frame: 6-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 8 | 9 | 9 | 10
score on a scale | 16.25 (6.67) | 20.78 (10.67) | 19.11 (10.43) | 20.20 (7.43)

21. Primary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Description: Patient-Reported Outcomes Measurement Information System (PROMIS-29) has seven categories: Physical Function (higher scores = better function), Anxiety (higher scores = more anxiety), Depression (higher scores = more depression), Fatigue (higher scores = more fatigue), Sleep Disturbance (higher scores = more disturbance during sleep), Pain (higher scores = more pain), and Social Function (higher scores = more socialization). Minimum score is 20 and maximum is 80 for each of the seven categories.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 11 | 11 | 12 | 12
score on a scale
  Anxiety | 46.96 (9.02) | 49.20 (8.29) | 53.81 (10.55) | 43.92 (5.99)
  Depression | 44.55 (6.09) | 41 (0) | 49.63 (11.19) | 43.88 (4.82)
  Fatigue | 53.49 (12.56) | 42.73 (6.92) | 49.33 (12.54) | 43.95 (6.78)
  Pain | 57.86 (6.32) | 53.65 (7.74) | 59.46 (7.31) | 56.69 (4.77)
  Sleep Disturbance | 52.35 (4.67) | 50.59 (8.91) | 54.44 (2.30) | 48.16 (8.55)
  Physical Function | 40.13 (4.36) | 46.52 (8.83) | 40.36 (6.19) | 44.32 (6.85)
  Social Function | 52.75 (8.96) | 53.27 (7.64) | 50.20 (9.06) | 54.99 (7.67)

22. Primary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Description: as for outcome 21
Time Frame: 3-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 12 | 10
score on a scale
  Anxiety | 47.54 (8.76) | 47.99 (8.38) | 52.88 (16.25) | 43.38 (6.22)
  Depression | 45.39 (6.50) | 43.12 (6.36) | 51.37 (13.63) | 43.59 (5.63)
  Fatigue | 48.90 (7.05) | 43.08 (10.13) | 49.92 (16.15) | 43.89 (8.29)
  Pain | 56.80 (3.68) | 50.93 (9.12) | 55.35 (7.37) | 53 (6.47)
  Sleep Disturbance | 50.58 (6.45) | 50.19 (8.25) | 52.48 (9.23) | 47.92 (7.77)
  Physical Function | 43.02 (5.78) | 49.35 (8.29) | 43.05 (7.02) | 48.36 (7.94)
  Social Function | 50.85 (6.03) | 54.56 (7.17) | 50.93 (7.93) | 56.12 (8.16)

23. Primary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Description: as for outcome 21
Time Frame: 6-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 9 | 11 | 10
score on a scale
  Anxiety | 43.30 (8.49) | 43.44 (6.08) | 53.60 (12.99) | 44.52 (7.11)
  Depression | 44.24 (6.82) | 44.07 (5.75) | 52.16 (13.81) | 43.92 (6.54)
  Fatigue | 49.86 (6.73) | 42.13 (8.75) | 49.05 (13.77) | 47.89 (9.72)
  Pain | 51.57 (6.30) | 50.84 (7.60) | 55.26 (7.51) | 51.21 (7.18)
  Sleep Disturbance | 49.27 (6.89) | 53.06 (8.19) | 49.96 (9.85) | 50.45 (3.60)
  Physical Function | 46.18 (6.97) | 48.34 (8.73) | 46.33 (5.80) | 46.73 (6.17)
  Social Function | 54.44 (8.12) | 53.00 (7.33) | 55.08 (10.09) | 54.02 (7.26)

24. Primary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Description: as for outcome 21
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 11 | 10
score on a scale
  Anxiety | 43.30 (8.49) | 46.59 (7.26) | 52.07 (10.44) | 43.18 (6.49)
  Depression | 43.94 (8.33) | 45.54 (5.95) | 50.04 (9.76) | 44.27 (7.53)
  Fatigue | 47.43 (7.48) | 46.16 (9.14) | 50.91 (11.42) | 46.74 (8.28)
  Pain | 48.56 (8.55) | 51.44 (8.99) | 53.72 (8.91) | 50.46 (8.04)
  Sleep Disturbance | 53.71 (4.37) | 50.51 (9.36) | 54.57 (3.82) | 51.71 (7.33)
  Physical Function | 49.71 (7.41) | 49.70 (9.32) | 45.27 (5.30) | 48.70 (5.81)
  Social Function | 54.26 (5.75) | 55.00 (8.17) | 52.36 (7.85) | 60.40 (4.98)

25. Primary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Description: as for outcome 21
Time Frame: 6-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 8 | 9 | 9 | 10
score on a scale
  Anxiety | 42.94 (6.98) | 45.47 (7.31) | 55.58 (14.81) | 43.95 (7.62)
  Depression | 43.24 (5.92) | 44.07 (5.75) | 49.96 (9.45) | 44.63 (7.85)
  Fatigue | 44.89 (7.97) | 44.87 (10.47) | 46.17 (14.26) | 40.42 (5.90)
  Pain | 52.46 (5.85) | 50.30 (10.43) | 52.63 (7.36) | 48.11 (7.24)
  Sleep Disturbance | 50.48 (7.53) | 50.90 (10.77) | 52.40 (11.16) | 50.49 (3.60)
  Physical Function | 49.79 (8.10) | 48.64 (9.43) | 46.46 (8.10) | 50.98 (6.56)
  Social Function | 53.86 (6.15) | 55.78 (9.69) | 52.27 (7.65) | 59.82 (6.58)

26. Primary Outcome: Cross-sectional Area
Description: Measures of interest include cross-sectional area. A study team member will assess ultrasound measures at baseline for both limbs, measured in centimeters (cm).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 11 | 11 | 12 | 12
Number analyzed (Limbs) | 22 | 22 | 24 | 24
cm | 0.64 (0.11) | 0.65 (0.15) | 0.69 (0.29) | 0.85 (0.27)

27. Primary Outcome: Cross-sectional Area
Description: Measures of interest include cross-sectional area. A study team member will assess ultrasound measures at 12 weeks for both limbs, measured in centimeters (cm).
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 11 | 10
Number analyzed (Limbs) | 18 | 20 | 22 | 20
cm | 0.67 (0.42) | 0.71 (0.21) | 0.62 (0.22) | 1.50 (1.39)

28. Primary Outcome: Cross Sectional Area
Description: Measures of interest include cross-sectional area. A study team member will assess ultrasound measures at 6 months for both limbs, measured in centimeters (cm).
Time Frame: 6-month
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 8 | 9 | 9 | 10
Number analyzed (Limbs) | 16 | 18 | 18 | 20
cm | 0.76 (0.38) | 0.74 (0.13) | 0.70 (0.33) | 0.80 (0.31)

29. Primary Outcome: Width
Description: Measures of interest include width of tendon. A study team member will assess ultrasound measures at baseline for both limbs, measured in centimeters (cm).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 11 | 11 | 12 | 12
Number analyzed (Limbs) | 22 | 22 | 24 | 24
cm | .563 (.10) | .59 (.13) | .59 (.31) | .69 (.16)

30. Primary Outcome: Width
Description: Measures of interest include width of tendon. A study team member will assess ultrasound measures at 12 weeks for both limbs, measured in centimeters (cm).
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 11 | 10
Number analyzed (Limbs) | 18 | 20 | 22 | 20
cm | .66 (.21) | .56 (.21) | .65 (.25) | .66 (.14)

31. Primary Outcome: Width
Description: Measures of interest include width of tendon. A study team member will assess ultrasound measures at 6 months for both limbs, measured in centimeters (cm).
Time Frame: 6-month
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 8 | 9 | 9 | 10
Number analyzed (Limbs) | 16 | 18 | 18 | 20
cm | .63 (.19) | .65 (.12) | .59 (.14) | .68 (.14)

32. Primary Outcome: Degree of Thickening
Description: Measures of interest include degree of thickening of tendon. A study team member will assess ultrasound measures at baseline for both limbs, measured in centimeters (cm).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 11 | 11 | 12 | 12
Number analyzed (Limbs) | 22 | 22 | 24 | 24
cm | 1.4 (.18) | 1.52 (.10) | 1.45 (.16) | 1.49 (.24)

33. Primary Outcome: Degree of Thickening
Description: Measures of interest include degree of thickening of tendon. A study team member will assess ultrasound measures at 12 weeks for both limbs, measured in centimeters (cm).
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 11 | 10
Number analyzed (Limbs) | 18 | 20 | 22 | 20
cm | 1.43 (.22) | 1.37 (.44) | 1.46 (.23) | 1.49 (.20)

34. Primary Outcome: Degree of Thickening
Description: Measures of interest include degree of thickening of tendon. A study team member will assess ultrasound measures at 6 months for both limbs, measured in centimeters (cm).
Time Frame: 6-month
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 8 | 9 | 9 | 10
Number analyzed (Limbs) | 16 | 18 | 18 | 20
cm | 1.45 (.24) | 1.53 (.17) | 1.37 (.13) | 1.55 (.25)

35. Primary Outcome: Relative Neovascularity
Description: Measures of interest include relative neovascularity. A study team member will assess ultrasound measures at baseline for both limbs. The relative level of neovascularization will be rated from grade 0: no visible vessels, grade 1: 1 to 2 vessels within the region of interest, grade 2: 3 to 5 vessels within the region of interest (ROI), or grade 3: vessel's in up to 30% of the ROI.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 11 | 11 | 12 | 12
Number analyzed (Limbs) | 22 | 22 | 24 | 24
score on a scale | .25 (.66) | .67 (.94) | .43 (.73) | 1.00 (1.15)

36. Primary Outcome: Relative Neovascularity
Description: Measures of interest include relative neovascularity. A study team member will assess ultrasound measures at 12 weeks for both limbs. The relative level of neovascularization will be rated from grade 0: no visible vessels, grade 1: 1 to 2 vessels within the region of interest, grade 2: 3 to 5 vessels within the region of interest (ROI), or grade 3: vessel's in up to 30% of the ROI.
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 11 | 10
Number analyzed (Limbs) | 18 | 20 | 22 | 20
score on a scale | .56 (1.07) | .89 (1.20) | .60 (.80) | 1.10 (1.30)

37. Primary Outcome: Relative Neovascularity
Description: Measures of interest include relative neovascularity. A study team member will assess ultrasound measures at 6 months for both limbs. The relative level of neovascularization will be rated from grade 0: no visible vessels, grade 2: 3 to 5 vessels within the region of interest (ROI), grade 3: vessel's in up to 30% of the ROI
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 8 | 9 | 9 | 10
Number analyzed (Limbs) | 16 | 18 | 18 | 20
score on a scale | .88 (1.27) | .56 (.83) | .89 (.99) | .60 (.92)

38. Primary Outcome: Elastography
Description: Measures of interest include elastography. A study team member will assess ultrasound measures at baseline for both limbs.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: m/s
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 11 | 11 | 12 | 12
Number analyzed (Limbs) | 22 | 22 | 24 | 24
m/s | 6.64 (.72) | 7.37 (.75) | 6.17 (.94) | 6.57 (.54)

39. Primary Outcome: Elastography
Description: Measures of interest include elastography. A study team member will assess ultrasound measures at 12 weeks for both limbs.
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: m/s
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 11 | 10
Number analyzed (Limbs) | 18 | 20 | 22 | 20
m/s | 6.70 (.66) | 6.63 (.70) | 6.40 (1.04) | 6.02 (.56)

40. Primary Outcome: Elastography
Description: Measures of interest include elastography. A study team member will assess ultrasound measures at 6 months for both limbs.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: m/s
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 8 | 9 | 9 | 10
Number analyzed (Limbs) | 16 | 18 | 18 | 20
m/s | 6.63 (.79) | 6.76 (.95) | 6.34 (.80) | 6.89 (.72)

41. Primary Outcome: Heel Raises-Quantitative Function in Heel Raises to Fatigue.
Description: Quantitative function in heel raises to fatigue on both limbs.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: heel raises
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 11 | 11 | 12 | 12
Number analyzed (Limbs) | 22 | 22 | 24 | 24
heel raises | 16.5 (8.62) | 15.50 (9.09) | 12.67 (7.63) | 15.73 (7.86)

42. Primary Outcome: Heel Raises-Quantitative Function in Heel Raises to Fatigue.
Description: Quantitative function in heel raises to fatigue on both limbs.
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: heel raises
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 11 | 10
Number analyzed (Limbs) | 18 | 20 | 22 | 20
heel raises | 28 (10.12) | 20.60 (7.63) | 21.80 (8.45) | 21.90 (6.09)

43. Primary Outcome: Heel Raises-Quantitative Function in Heel Raises to Fatigue.
Description: Quantitative function in heel raises to fatigue on both limbs.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: heel raises
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 8 | 9 | 9 | 10
Number analyzed (Limbs) | 16 | 18 | 18 | 20
heel raises | 22.13 (5.56) | 21.44 (6.96) | 20.22 (4.13) | 21.90 (10.52)

44. Primary Outcome: Hops
Description: Quantitative function in ankle strength, we will also ask the participants to complete 20 hops and rate their pain using the Defense and Veteran's Pain Rating Scale (DVPRS). The Defense and Veterans Pain Rating Scale (DVPRS) is a pain assessment tool designed specifically for military personnel and veterans Rating scale from 0-10. Higher scores equal worse outcomes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 11 | 11 | 12 | 12
score on a scale | 3.18 (2.21) | 3.20 (2.71) | 4.92 (3.15) | 2.70 (1.85)

45. Primary Outcome: Hops
Description: as for outcome 44
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 11 | 10
score on a scale | .44 (.68) | 2.40 (1.85) | 3.20 (2.44) | 1.90 (1.45)

46. Primary Outcome: Hops
Description: as for outcome 44
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 8 | 9 | 9 | 10
score on a scale | .88 (1.69) | 2.38 (2.91) | 3.00 (2.11) | 2.10 (2.88)

47. Primary Outcome: Ankle Range of Motion (ROM)
Description: Quantitative function in range of motion (ROM).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 11 | 11 | 12 | 12
Number analyzed (Limbs) | 22 | 22 | 24 | 24
degrees | 12.18 (4.39) | 12.40 (4.18) | 12.67 (9.74) | 12.18 (4.04)

48. Primary Outcome: Ankle Range of Motion (ROM)
Description: Quantitative function in range of motion (ROM)
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 9 | 10 | 11 | 10
Number analyzed (Limbs) | 18 | 20 | 22 | 20
degrees | 14.89 (3.14) | 13.80 (6.29) | 10.60 (3.58) | 10.80 (3.37)

49. Primary Outcome: Ankle Range of Motion (ROM)
Description: Quantitative function in range of motion (ROM)
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Limbs
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
Number analyzed (Participants) | 8 | 9 | 9 | 10
Number analyzed (Limbs) | 16 | 18 | 18 | 20
degrees | 15.75 (7.64) | 10.22 (3.46) | 10.67 (4.32) | 11.60 (5.12)

ADVERSE EVENTS:
Time Frame: All participants were evaluated for adverse events at each follow-up visit during their participation in the study (at 3 weeks, 6 weeks, 3 months, and 6 months), and all reportable events, regardless of severity, were reported to the Principal Investigator and the IRB.
Description: The study overall is considered to be minimal risk for study participants: not substantially above what would be encountered in everyday life including provision of routine medical care for the condition of Achilles tendinopathy.
  All reportable events, regardless of severity, were reported to the Principal Investigator and the Institutional Review Board. All adverse events were reviewed and made a determination of severity and relationship to participation in the research study.
Groups:
- Physical Therapy (PT) Only: In Part 1, the physical therapy only arm requires 8 visits. The participants will complete 2 check-in visits each week (remote or in person), for three weeks. Follow-up data will be collected at 6 weeks (virtual or in-person) and at 3 months (in-person).
  Physical Therapy: All participants may complete a PT program as standard of care (SOC) treatment addressing individual strength, mobility, and flexibility deficits in both proximal (e.g. spine and hip girdle) along with distal (thigh, leg, and foot/ankle) muscle groups. The provider may also use other modalities to address distal issues. To standardize the loading program, all participants will be given an at-home exercise program designed by Dr. Karin Sibernagel for progressive Achilles tendon loading. The participants will also follow the University of Delaware Return to Sport protocol for return to running. This will be completed alongside the standard of care PT participants will be receiving.
- PT + SWT and PBMT: The PT + SWT + PBMT arm will receive both SWT and PBMT treatments in addition to PT treatment described. Participants will receive PBMT twice a week and SWT once a week, for three weeks. The SWT visit may be combined with a PBMT visit in the same week. Up to two times each week after a treatment visit (for three weeks), a team member will check-in with the participants to ensure physical therapy exercise adherence, and response to treatment. During the second check-in of the week, the team member will also ensure the participant is keeping their activity/medication/pain log; the team member will also deliver the DVPRS with supplemental questions. When/if needed, these check-ins may occur virtually. (See Appendix F for check-in data collection CRF).
Arm/Group | Physical Therapy (PT) Only | PT + Photobiomodulation Therapy (PBMT) | PT + Shockwave Therapy (SWT) | PT + SWT and PBMT
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 4/11 | 2/10 | 2/12 | 0/12
Other Adverse Events (participants affected / at risk) | 8/11 | 8/10 | 9/12 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Therapy (PT) Only (N=11) | PT + Photobiomodulation Therapy (PBMT) (N=10) | PT + Shockwave Therapy (SWT) (N=12) | PT + SWT and PBMT (N=12)
Shoulder Surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant had right shoulder surgery. Not related to the research procedures.
Neck Surgery (Surgical and medical procedures) | 0 | 1 (1) | 0 (0) | 0 (0) — Participant had a spinal neck surgery. Not related with the study procedures.
URI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant went to Emergency Department for URI. Not related to study procedures.
Achilles Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant went to ER for Bilateral Achilles pain. Aggravated after walking for hours and got an anti-inflammatory injection for the pain.
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant went to hospital for rhabdomyolysis. Not related to the study procedures.
Allergy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — participant went to Emergency Department due to skin reaction from laundry detergent.
Sprained Ankle (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Ankle sprained. Injury was treated.
Emergency Department (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported visiting emergency department; detail is unknown.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Therapy (PT) Only (N=11) | PT + Photobiomodulation Therapy (PBMT) (N=10) | PT + Shockwave Therapy (SWT) (N=12) | PT + SWT and PBMT (N=12)
Achilles Pain in non-study leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Achilles Pain in non-study leg.
Cervical Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant reported consult appointment for cervical pain and possible surgery. Not related to the study.
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Flare up of right knee gout symptoms. Not related to the study procedures.
Heel Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant reported new heel pain on right side of the foot. Not related to the study procedures.
Pain in Achilles (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant reported pain in Achilles, stiff in morning. Relives with at-home exercises.
Knee Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Injured left knee while playing football. Not related to the study procedures.
Aggravated Achilles (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Aggravated right Achilles more than usual.
Food poison (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Had food poisoning and was fine after rest. Not related to study procedures.
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — Participant experienced shoulder pain. Being treated conservatively and seeing PT for it. Not related to the study procedures.
Foot and Achilles Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant reported Right Foot soreness and left Achilles soreness.
Increased Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Pain in back of both knees. After doing study exercises, the pain lingering for a few days.
Sore Calf (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Increased left calf soreness.
Running increases Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant reported a slight increase in pain when running.
Cortisone Injection (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant had cortisone injection on shoulder. Not related to study procedures.
Aggravated Achilles (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Aggravated right achilleas more than usual. Not related to the study procedures.
Increased soreness from standing (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant reported increased soreness from Stading at work. Symptoms resolved.
Increased soreness in Achilles (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Increased soreness in the Achilles.
Plantar fascia in non-study leg (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Participant reported pain in non-study leg plantar fascia. Being treated at PT. Not related to the study procedures.
Increased Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant reported worsening of pain over week-2, maximum pain during ACFT.
Left Knee Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Knee injury while working out. Not related to the study.
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Injured while playing soccer. Calf sore increased.
Treatment for Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant reported pain and took Diclofenac for left hallux. Not related to study procedures.
Increased Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Increased pain when trying to run half mile. Rested and feeling back to baseline.
Increased Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant reported noticing increased Pain with new boots.
Increased Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant reported feeling increased in symptoms in their Achilles region while they were cooking in the kitchen and turned awkwardly. The symptoms were resolved withing 24 hours which is to be expected during the healing phase following an injury.
Increased Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Noted increased pain while sprinting. Symptoms reduced over the weekend.
Increased Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant reported increased in pain while sleeping. Rested several days and reported feeling better.
Increased Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Noted increased left Achilles pain. Has moved towards the inside.
Increased left Achilles Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Increased pain in left achilles post at home exercise. 3 pain reduces to 0 an hour post exercise.
Increased Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant reported feeling increased soreness when walking. Improved with rest.
Increased Achilles Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Increased Achilles pain. Symptoms subsided with within 48 hours.
Achilles Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Pain with movement in left Achilles after shockwave therapy. Continued to monitor and pain has subsided.
Ankle Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant was noting an increase in left ankle soreness and symptoms during home exercise program. The symptom resolved within 2 days which is to be expected with the initiation of a home exercise program.
Injection in the eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant reported receiving the Beovu injection in the right eye and followed up with by ophthalmology department. Not related to the study procedures.
Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant reported that they felt more sore than usual after doing exercises day before.
Soreness, tenderness, and stiffness in a Achilles (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant reported having soreness, tenderness, and stiffness as expected from exercises. Participant also reported have more symptoms at night.
Increased Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant reported soreness increased after walking over the weekend.
Increased Achilles Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Increased Achilles pain while on TDY. No MOI.
Increased Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant reported feeling increased in pain while moving out over the weekend.
Soreness in Calf (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Increased soreness in the calf.
Increased Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Increased soreness in the calf.
Slight increase in Achilles symptoms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant reported feeling slight increases in Achilles symptoms with exercises.
Hamstring Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant reported injuring hamstring from playing soccer. Not related to the study procedures
Tightness in Achilles (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Notes the Achilles was tight while playing soccer over the weekend and loosened up with some stretching.
Increase in Achilles Symptoms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant notes an increase in symptoms in Achilles several weeks ago. Insidious onset and since the increase in pain, symptoms are improving. Continue to monitor and reassess.
Pain in Achilles (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported pain in Achilles after 3-mile run, iced area.
Pain in Achilles (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pain in right Achilles day after Shockwave therapy, was at range all day. Pain resolved in 48 hours.
Pain in Non-Study Foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported pain in non-study(left) Achilles that wasn't present before.
Emergency Department (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported that they went to emergency department, detail is unknown.
Pain in Achilles (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pain in Achilles post-run following into the next am: resting. continue to monitor.
Worsening of Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pain worsened after trying to sprint. Treated clinically and able to progress. Will monitor.
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported that they went to Primary Care Provider for a cough. Had an elevated blood pressure reading.
Teeth Extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported that they had a wisdom teeth extraction.
Pain in Non-study Achilles (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported that they experienced new pain in non-study Achilles after training; is lingering; will monitor.
Lingering Pain in Achilles (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported that the pain in their left Achilles is lingering days after Shockwave therapy. Will monitor and evaluate at next Shockwave therapy appointment.
Increased Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Increased soreness during heel raises. Modifying reps.
Increased Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported that they felt increased soreness. Trying to rub. Will follow-up to see progression.
Increased Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported that they felt increased soreness. Loosened up as the day progressed. Participant did not report continued symptoms.
Pain and Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported pain at Achilles and a bit sore when working.
Increased Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported experiencing increased soreness in the Achilles region while performing heel raise exercise. The symptoms were minimal in presentation and not unexpected following start of a loading program for the Achilles tendon.
Calf Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported increasing in calf soreness. Achilles is feeling better.
Achilles Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported they slipped while weight lifting which caused the left ankle and Achilles soreness.
Neck and Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant reported seeing Physical Therapist and Chiropractor for their neck and back. Not related to the study procedures.
Tingling Sensation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant reported tingling sensation when rolling study ankle, shoots down ankle to foot. Started after hop test.
Heel Issue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant reported feeling issues with bottom of heel when doing heel raises.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT05751785/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT05751785/ICF_001.pdf